CLINICAL TRIAL: NCT01692327
Title: Evaluating the Effect of Lipid Overload in Endothelial Function and Microvascular Reactivity in Young Obese Women
Brief Title: Study About High Fat Meal and Postprandial Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Priscila Alves Maranhao, Nutricionist, Rio de Janeiro State University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Biovasc-02; Biovasc002 (Registry Identifier: Over load project)
Record Dates: First submitted 2012-09-12; First posted 2012-09-25 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: glucose intolerance (20); Control (20)
MeSH Terms: conditions — Obesity; Glucose Intolerance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Obese Group (Other): Obese group with fat overload intake.
  Interventions: Dietary Supplement: High fat meal
- Control Group (Other): Control Group + fat overload intake
  Interventions: Dietary Supplement: High fat meal
- Glucose Intolerance (Other): glucose intolerance + fat overload intake
  Interventions: Dietary Supplement: High fat meal

INTERVENTIONS:
Dietary Supplement: High fat meal

SUMMARY:
The hypothesis of the proposed project is that after a fat overload, the postprandial response is different in both groups, suggesting that the LPP will present the most significant damage in endothelial vasomotion in obese individuals, especially those with GI and T2DM. After the fat overload, we hypothesized that there will be a worsening of endothelial function and microvascular reactivity in OB/DM2 and OB group compared to C, but also find lower concentrations of incretins in OB/DM2 group compared to other groups.

These hypotheses may be confirmed by techniques for evaluating microvascular function, the use of DFT skin for vasomotion evaluation and finally analysis of analytes through metabolic and cardiovascular read by Multiplex kit.

DETAILED DESCRIPTION:
Will be recruited 60 women aged 19-40 years, with a diagnosis of obesity (BMI ≥ 30 kg/m2) treated at the obesity clinic at the State University of Rio de Janeiro (UERJ)at Brazil.

Microcirculation parameters and blood tests will be assessed at baseline and after this, the women will receive a high-fat meal containing croissant, salami, whole milk and cheddar cheese. After 30, 60, 120 and 180 minutes this meal the microcirculation will be evaluated as well as blood collection.

ELIGIBILITY:
Inclusion Criteria:

* all patients should have obesity class I (BMI between 30 and 35kg/m2);
* Submit diabetes mellitus without further treatment or be obese non-diabetic or glucose intolerant;
* Presenting the age between 19 to 40 years.
* Waist circumference> 80 cm (IDF)

Exclusion Criteria:

* Renal disease, coronary or peripheral vascular, hematologic or hepatic impairment;
* Presence of dyslipidemia;
* smokers;
* Significant loss of body weight six months prior to the study.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Microvascular function | up to 180 minutes after high fat meal

SECONDARY OUTCOMES:
incretins hormones | basal, 30, 60, 120,180 minutes after high fat meal
  We will assess incretins hormones by multiplex

CONTACTS AND LOCATIONS:
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] de Souza MDGC, Maranhao PA, Panazzolo DG, Nogueira Neto JF, Bouskela E, Kraemer-Aguiar LG. Effects of a high-fat meal on inflammatory and endothelial injury biomarkers in accordance with adiposity status: a cross-sectional study. Nutr J. 2022 Oct 19;21(1):65. doi: 10.1186/s12937-022-00819-4. PMID 36258233